CLINICAL TRIAL: NCT07039448
Title: Effectiveness of Self-Administered Acupressure Intervention in Managing Constipation of Adult Psychiatric In-Patient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr Kelvin WONG Wai Kit, Assistant Professor, School of Nursing and Health Sciences, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2024-301
Record Dates: First submitted 2025-06-02; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Constipation; Psychiatric Drug Induced Constipation; Constipation Drug Induced
Keywords: constipation; psychiatric in-patient
MeSH Terms: conditions — Constipation | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The acupressure intervention including the five acupoints are Zhongwan (RN12), which are located on the upper abdomen and on the anterior midline 4 cun (just over 10 cm) above the center of the umbilicus; the right and left Tianshu (ST25), located in the central abdominal region and 2 cun (just over 5 cm) lateral to the umbilicus; and the right and left Quchi (LI11), located at the lateral end of the transverse elbow crease when the forearm is flexed and at the midpoint of the line connecting Chize (LU5) to the lateral epicondyle of the humerus. The acupressure will be performed once a day for 10 days in a group setting with same sex, supervised by a trained psychiatric nurse and preferably at least 2 hours after a meal.
  Interventions: Behavioral: Acupressure
- Sham Control Group (Sham Comparator): The sham group will be trained to perform acupressure in a similar way to the intervention group, except that they will use five sham acupoints. After completion of the project, patients in the sham group will receive the same interventions as the intervention group.
  Interventions: Behavioral: Sham Comparator

INTERVENTIONS:
Behavioral: Acupressure — The acupressure intervention including the five acupoints. The acupressure will be performed once a day for 10 days in a group setting with same sex, supervised by a trained psychiatric nurse and preferably at least 2 hours after a meal.
  Arms: Treatment Group
Behavioral: Sham Comparator — The sham group will be trained to perform acupressure in a similar way to the intervention group, except that they will use five sham acupoints. After completion of the project, patients in the sham group will receive the same interventions as the intervention group.
  Arms: Sham Control Group

SUMMARY:
Constipation is a common gastrointestinal condition characterized by unsatisfactory defaecation as a result of infrequent stools, difficult stool passage, or both. Overall, the average prevalence of constipation was estimated at 16% worldwide. It affects about 14.3% of the population in Hong Kong. The condition incurs significant costs, with over £162 million in the UK National Health Service from 2017 to 2018. Similar high expenses are reported in Hong Kong and many Western countries. Studies have shown that constipation can lead to serious health complications, including paralytic ileus, fecal impaction, bowel obstruction, and even premature death. It not only causes patient discomfort and reduces quality of life, but also increases treatment costs.

Psychiatric patients, particularly those on psychotropic drugs such as antipsychotics and antidepressants, are more susceptible to constipation, with over a third affected in Europe. This high prevalence may be due to the side effects of antipsychotics and antidepressant drugs, as well as factors like limited physical activity, sedentary lifestyle, negative symptoms, poor mental state, unhealthy diet, and insufficient fiber intake. The physical health of individuals with severe mental illness, including constipation, has become a major concern in recent years. However, these issues are often overlooked and under-researched, making its management a critical aspect of mental health care.

Common treatments of constipation include pharmacological and non-pharmacological interventions. While pharmacological intervention can effectively alleviate symptoms, it is a short-term solution but long-term use of laxatives can cause serious side effects such as bloating, allergic reaction, abdominal pain, metabolic disturbances, and hepatotoxicity that can far outweigh the therapeutic effects of symptom reduction. Alternative non-traumatic interventions like auriculotherapy and behavioral therapy have been found to be ineffective. Only one RCT study of abdominal massage therapy to 60 elderlies with constipation in Sweden has shown decrease severity of constipation and increased bowel movement but did not lead to decrease in laxative intake, also the intervention requires a therapist to perform. This may reduce the accessibility and sustainability of the intervention to manage constipation. Therefore, the investigators propose to test a simpler and less expensive intervention to manage constipation to adult psychiatric patient. This intervention incorporates the concept of self-help, acupressure into the project.

Self-help concept: Since the 19th century, self-care has been a crucial element within healthcare systems. It is characterized as a deliberate action undertaken by an individual to enhance health or manage disease. Florence Nightingale underscored the significance of personal hygiene and environmental factors in health, thereby establishing self-care as a fundamental principle in public health nursing. Orem further developed the notion of self-care, classifying it into three categories: universal self-care requisites, developmental self-care requisites, and health-deviation self-care requisites. Barofsky divided self-care activities into four types: regulatory, preventive, reactive, and restorative self-care. Both the World Health Organization and Pender accentuated the function of self-care in health enhancement, disease prevention, and health restoration. In Orem's self-care model, nursing therapeutics are divided into five categories, with patients perceived as active contributors to their own care.

Acupressure: Acupressure involves the application of constant pressure by fingertip, thumb or palm to specific acupoints for stimulating the flow of 'Qi' in the meridians. In TCM, health problems are deemed to be due to pathogenic changes in 'Qi' and imbalance of 'Yin' and 'Yang'. Dysfunction of the viscera and bowels is induced by a deficiency or excess of 'Qi' in the body. The acupressure is based on the Meridian theory that a life force called 'Qi' flows through the body along certain channels (meridians), which if blocked can cause illness. Stimulation at precise locations (acupoints) along these channels by healthcare provider or patients themselves can unblock the flow of 'Qi', relieving pain and restoring health. Acupressure is able to influence autonomic functions, which can affect the functioning of defecation. In addition, Some studies found that acupressure improved symptoms of constipation in elderly, stroke, and vegetative status patients. Acupressure might have positive effect of improving constipation in patients. Unfortunately, there is no trails (RCT or non-RCT) on psychiatric patient. Therefore this intervention will be tested among the psychiatric in-patients in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong Chinese residents, aged 18 or above
2. Meet the diagnostic criteria of Rome III for constipation
3. Mentally stable and competent for self-care and learning acupressure, as recommended by their attending psychiatrists and
4. Able to understand the questionnaire and follow instructions for training will be eligible to participate in this study

Exclusion Criteria:

1. Anatomical and physiological disorders of gastrointestinal tract such as malrotation, fistula and colonic neuropathies
2. Metabolic and endocrine diseases
3. Lead poisoning and vitamin D intoxication
4. Previous training in acupressure
5. Physical disability involved the upper limbs
6. Planned surgery undergoing during study period and pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Severity of constipation symptoms | Pre-intervention, Immediately after intervention, 4-weeks after post-intervention, 8-week after post-intervention
  Chinese version of Constipation Assessment Scale (C-CAS) will be used to assess the severity of constipation symptom: The 8-item C-CAS has been commonly used with 3-point Likert scale, including '0= no problem', '1= some problem', and '2= severe problem'.
Number of Complete Spontaneous Bowel Movements | Pre-intervention, Immediately after intervention, 4-weeks after post-intervention, 8-week after post-intervention
  The number of Complete Spontaneous Bowel Movements (CSBM) will be used to measure symptom severity of constipation which is recorded in the Patient's Bowel Movement Chart (MR402351/NTWC).
Stool form | Pre-intervention, Immediately after intervention, 4-weeks after post-intervention, 8-week after post-intervention
  Bristol Stool Form Scale (BSFS) will be used to measure symptom severity of constipation. The Bristol Stool Form Scale (BSFS), a graded visual scale of stool type from type 1 (hard lumps) to type 7 (watery diarrhea) which is recorded in the Patient's Bowel Movement Chart (MR402351/NTWC), will be used to assess the patient's stool form.
Use of medication to relieve constipation symptoms | Pre-intervention, Immediately after intervention, 4-weeks after post-intervention, 8-week after post-intervention
  The reduction of using medication to to relive constipation symptoms

SECONDARY OUTCOMES:
Patient's quality of life | Pre-intervention, Immediately after intervention, 4-weeks after post-intervention, 8-week after post-intervention
  Chinese version of Patient Assessment Constipation Quality of Life Questionnaire (C-PAC-QoL) will be used to assess the specific disease related patient quality of life: The PAC-QoL consists of 28 items categorised into four subscales, including dissatisfaction (5 items), physical discomfort (4 items), psychosocial discomfort (8 items), and worries and concerns (11 items) with 5-point Likert scale, ranging from '0 = none of the time or not at all' to '4 = all of the time or extremely'. The lower average total score indicates the better the person's health-related quality of life.

OTHER OUTCOMES:
Participants' perceptions of the benefits of the intervention | 8-weeks after post-intervention
  Focus group will be held with participants to discuss the perceptions of the benefits of the intervention experienced, any positive effects in reducing constipation and its related suffering, and any difficulties encountered during the intervention
Nurses' perceptions of the intervention | 8-weeks after post-intervention
  Focus group will be held with research nurses on the feedback and comments on the adequacy and feasibility of the content and procedure of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Peak Hospital, Tuenmen, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No